CLINICAL TRIAL: NCT03823508
Title: Prefontal tDCS in Patients With Disorders of Consciousness: Neurophysiological and Behavioural Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Aurore Thibaut, Principal Investigator, University of Liege
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-296
Record Dates: First submitted 2019-01-29; First posted 2019-01-30 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Vegetative State; Minimally Conscious State; Disorder of Consciousness
Keywords: Vegetative state; Minimally Conscious State; Disorders of consciousness; Transcranial direct current stimulation; Non invasive brain stimulation; Neuromodulation; High density electroencephalography
MeSH Terms: conditions — Persistent Vegetative State; Consciousness Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anodal tDCS (Active Comparator): Patients will receive anodal tDCS (left dorsolateral prefrontal stimulation) during 20 minutes preceded and followed by a clinical assessment (Coma Recovery Scale-Revised) and neurophysiological assessment (256 channels EEG).
  Interventions: Device: anodal tDCS
- sham tDCS (Placebo Comparator): Patients will receive sham tDCS (15 secondes of stimulation) during 20 minutes preceded and followed by a clinical assessment (Coma Recovery Scale-Revised) and neurophysiological assessment (256 channels EEG).
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: anodal tDCS — Patients will receive anodal tDCS during 20 minutes preceded and followed by a behavioral assessment (Coma Recovery Scale Revised) and a high density EEG. The anode will be placed over F3 in order to stimulate the left dorsolateral prefrontal cortex and the cathode over the right supraorbital area.
  Arms: anodal tDCS
Device: sham tDCS — Identical to anodal tDCS, except that the stimulation will be stopped after 15 seconds.
  Arms: sham tDCS

SUMMARY:
Non-invasive brain stimulations techniques have recently shown promising results in patients with disorders. Notably, transcranial direct current stimulation (tDCS) applied over the left dorsolateral prefrontal cortex has proved to be effective in improving signs of consciousness in about 50% of patients in MCS either after a single stimulation or after repeated sessions. However, brain mechanisms underlying tDCS effects remain poorly understood. Here we aim to assess the effects of prefrontal tDCS on neurophysiological (i.e., electroencephalography - EEG - primary outcome) and behavioral (secondary outcome) measures in severely brain-injured patients with DOC.

DETAILED DESCRIPTION:
Currently, therapeutic options for severely brain-injured patients with disorders of consciousness (DOC), including patients in unresponsive wakefulness syndrome (UWS) and minimally conscious state (MCS), are limited and still need to be improved to influence long-term outcomes. Non-invasive brain stimulations (NIBS) techniques have recently shown promising results in DOC. Notably, transcranial direct current stimulation (tDCS) applied over the left dorsolateral prefrontal cortex has proved to be effective in improving signs of consciousness in about 50% of patients in MCS either after a single stimulation or after repeated sessions. However, brain mechanisms underlying tDCS effects remain poorly understood.In the present protocol, the investigators will assess the effects of prefrontal tDCS on neurophysiological (i.e., electroencephalography - EEG - primary outcome) and behavioral (secondary outcome) measures in severely brain-injured patients with DOC in a double-blind sham-controlled design. One anodal and one sham tDCS will be delivered in a randomized order in chronic (>28 days post-onset) severely brain-damaged patients. The stimulation will have an intensity of 2 mA and will last 20 minutes. The anode will be placed on the left dorsolateral prefrontal cortex and the cathode on the right supraorbital region. Ten minutes of high-density EEG will be recorded using a 256-channel saline electrode net (Electrical Geodesics) directly before and after each tDCS session. Behavioral assessments will be performed using the Coma Recovery Scale-Revised before and after each session by an investigator blinded to the treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

* post-comatose patients
* patients in vegetative state/unresponsive wakefulness syndrome or in minimally conscious state
* patients with stable condition
* patients free of sedative drugs and Na+ or Ca++ blockers (e.g., carbamazepine) or NMDA receptor antagonist (e.g., dextromethorphan)

Exclusion Criteria:

* premorbid neurology antecedent
* patients in coma
* patients < 28 days after the acute brain injury
* patients with a metallic cerebral implant/a shunt
* cranioplasty

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Change in the CRS-R scores | Baseline and directly after the tDCS (20 minutes)
  CRS-R will be performed before and after tDCS (anodal and sham). Comparison of the treatment effect (CRS-R total score after tDCS minus before) between real and sham tDCS

SECONDARY OUTCOMES:
Change in EEG | Baseline and directly after the tDCS (20 minutes)
  256 channels EEG will be record before and after tDCS to record potential cortical changes induce by the stimulation.
Change in the vigilance level | Baseline and directly after the tDCS (20 minutes)
  Ocular parameters will be record using glasses before and after tDCS to record potential change of the vigilance level

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Liege, Liège, Belgium